CLINICAL TRIAL: NCT03946553
Title: The Dysbiosis of the Intestinal Microbiota in Individuals With Allergic Rhinitis: an Observational Study (MICRORIN)
Brief Title: The Dysbiosis of the Intestinal Microbiota in Individuals With Allergic Rhinitis (MICRORIN)
Acronym: MICRORIN
Status: Completed | Type: Observational
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: Technological Centre of Nutrition and Health (Other); Biopolis S.L. (Industry); Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Sponsor
Other Study IDs: MICRORIN
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis
Keywords: intestinal microbiota; immunological markers
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allergic Rhinitis Group: Individuals with allergic rhinitis
- Control Group: Individuals without allergic rhinitis

INTERVENTIONS:
Other:  — No intervention
  Groups: Allergic Rhinitis Group

SUMMARY:
Allergic rhinitis (AR) is triggered by environmental allergens such as pollen and mites, and is associated with several symptoms such as itching and nasal congestion, sneezing or tearing and redness of the eyes. RA can affect patients life quality who suffer it, reducing the quality of sleep and cognitive function, causing irritability and fatigue and, consequently a decrease in work performance.

Because the existing pharmacological treatments for RA are not entirely effective, it is of interest to find other means to enhance the effects of these drugs and decrease more effectively the signs and symptoms associated with RA. In this context, RA has been related to an alteration of the intestinal microbiota (MI).However, there is a need to characterize in detail the MI of individuals who suffer RA.

The main objective of the present study is to characterize the MI of individuals with RA, compared with people without RA. In addition, the secondary objective is to study the association between characteristics of the MI of individuals with RA and different immunological markers.

ELIGIBILITY:
Inclusion Criteria Allergic Rhinitis population:

1. Men and women over 18 years of age.
2. Sign the informed consent.
3. Present, according to the ARIA classification (Allergic Rhinitis ans its impact on

   Asthma), two or more of the following symptoms for more than one hour a day:
   * Aqueous rhinorrhea.
   * Sneezing, especially paroxysmal.
   * Nasal obstruction.
   * Itching or nasal itch.
   * Conjunctivitis (itching, lacrimation or redness).
4. Individuals presenting Persistent or Perennial type of RA, in which signs are present:

   * More than four days a week.
   * And for more than four consecutive weeks.

Exclusion Criteria Allergic Rhinitis population:

1. Purulent Rhinorrhea.
2. Being pregnant.
3. Be in breastfeeding period.
4. Having diabetes (glucose ≥ 126 mg/dL).
5. BMI values > 30 kg/m^2.
6. Present dyslipidemia (LDL cholesterol ≥ 189 mg/dL and/or triglycerides ≥ 350 mg/dL).
7. Systolic Blood Pressure ≥ 160 mmHg and/or Diastolic Blood Pressure ≥ 100 mmHg.
8. Have received treatment with antibiotics 30 days before the start of the study.
9. Have received treatment with corticosteroids 30 days before the start of the study.
10. Individuals who usually intake prebiotics and/or probiotics supplements 30 days before the start of the study.

Inclusion Criteria Control population:

1. Men and women over 18 years of age.
2. Sign the informed consent.
3. Do not present any signs or symptoms of RA.

Exclusion Criteria Control population:

1. Being pregnant.
2. Be in breastfeeding period.
3. Having diabetes (glucose ≥ 126 mg/dL).
4. BMI values > 30 kg/m^2.
5. Present dyslipidemia (LDL cholesterol ≥ 189 mg/dL and/or triglycerides ≥ 350 mg/dL).
6. Systolic Blood Pressure ≥ 160 mmHg and/or Diastolic Blood Pressure ≥ 100 mmHg.
7. Have received treatment with antibiotics 30 days before the start of the study.
8. Have received treatment with corticosteroids 30 days before the start of the study.
9. Individuals who usually intake prebiotics and/or probiotics supplements 30 days before the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the study will be two types of populations. A population with allergic rhinitis and a population without allergic rhinitis and that serves as control group.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Intestinal microbiota characterization | At Day 1
  Taxonomic identification of the intestinal microbiota of the participants by sequencing the fecal DNA samples using MiSeq platform of Illumina in combination with 250/300PE.

SECONDARY OUTCOMES:
Inflammatory markers in blood | At Day 1
  Quantification of the pro-inflammatory markers Interleuquin (IL)-6 and TNFalpha and of the anti-inflammatory marker IL-10 in blood by ELISA kits.
Immunological markers in faeces | At Day 1.
  Quantification of Immunoglobulin (Ig) A levels in faeces by ELISA kit as a marker of intestinal inflammatory response.
Immunological markers in blood | At Day 1.
  Quantification of IgE by Phadiatop adults.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Dr, Principal Investigator — UTNS (Eurecat_Reus)/HUSJR. Reus, Tarragona, Spain.
Locations (1):
- Technological Centre of Nutrition and Health (Eurecat-Reus), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org
- See also: Biopolis S.L. — http://biopolis.es